CLINICAL TRIAL: NCT01091961
Title: Pre-Operative Inhibition of the Angiotensin System Study: A Prospective Randomized Single-Blinded Trial of Pre-Operative Management of Medications That Inhibit the Renin-Angiotensin System
Brief Title: Study of Preoperative Management of Angiotensin Converting Enzyme Inhibitor (ACEi) and Angiotensin Receptor Blocker (ARB) Medications
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-09-487; 16503 (Other: REB)
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Hypertension
Keywords: ACE inhibitor; ARB; Non-cardiac surgery; Perioperative; Preoperative; Hypotension; Congestive heart failure; Hypertension; Angiotensin-Converting Enzyme Inhibitors; Angiotensin II Type 1 Receptor Blockers; Perioperative Care
MeSH Terms: conditions — Hypertension; Hypotension; Heart Failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuing ACEi/ARB (Active Comparator): Patients in this group will continue to take their chronic ACEi/ARB medications up to and including the day of surgery.
  Interventions: Procedure: Preoperative ACEi/ARB management
- Holding ACEi/ARB (Active Comparator): Patients in this arm will hold their chronic ACEi/ARB medication at least 24 hours prior to surgery.
  Interventions: Procedure: Preoperative ACEi/ARB management

INTERVENTIONS:
Procedure: Preoperative ACEi/ARB management — Patients will either hold their chronic ACEi/ARB medication for at least 24 hours prior to surgery, or continue to take the ACEi/ARB medication up to and including the day of surgery

SUMMARY:
Patients on a stable dose of ACE inhibitor or ARB medication who are scheduled for elective surgery will be randomized to take their ACE inhibitor or ARB up to and including the morning of surgery, or to hold them a day prior to the surgery. The patients will be followed for 30 days after surgery to assess any adverse health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* currently taking an ACEi, ARB or both
* no change in these medications during the two weeks prior to study enrollment
* scheduled for non-cardiac surgery requiring regional or general anesthesia
* minimum overnight anticipated length of stay
* age ≥18 years.

Exclusion Criteria:

* explicit instructions provided to patient by surgical team regarding the perioperative management of ACEi or ARB
* significant hypertension in pre-operative assessment clinic (systolic blood pressure ≥180 mmHg OR diastolic blood pressure ≥110 mmHg)
* significant hypotension in pre-operative assessment clinic (systolic blood pressure < 90 mmHg)
* prior enrollment in the study
* participation in another research study of antihypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood pressure | 24 hours after surgery

SECONDARY OUTCOMES:
Clinically significant hypotension | 30 days after surgery
Clinically significant hypertension | 30 days after surgery
All-cause mortality | 30 days after surgery
Cardiovascular morbidity | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marko Mrkobrada, MD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada